CLINICAL TRIAL: NCT05188222
Title: The Effect of Preoperative Maltodextrin on Cardiac Function in Cardiac Surgery Patients with Reduced Left Ventricular Ejection Fraction: a Randomized, Controlled, Double-blind, Clinical Trial
Brief Title: Preoperative Maltodextrin's Effect on Cardiac Function in Cardiac Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Matthew Cameron, MDCM MPH, Assistant Professor, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MP-05-2022-3112
Record Dates: First submitted 2021-12-21; First posted 2022-01-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-09

CONDITIONS: Left Ventricular Dysfunction; Quality of Recovery; Right Ventricular Dysfunction
Keywords: Cardiac surgery; Insulin; Maltodextrin; Enhanced Recovery After Surgery; Quality of Recovery After Surgery
MeSH Terms: conditions — Ventricular Dysfunction, Left; Ventricular Dysfunction, Right; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to the intervention or control group based on a computer-generated 1:1 stratified block randomization by procedure type in blocks of 4, stratified by sex.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Packets of the study drug will be prepared by Enhanced Medical Nutrition and look identical. The placebo has been formulated to taste the same as Maltodextrin as well
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group will receive an oral preparation of 50 grams of Maltodextrin solution mixed in 400 millilitres (mL) of water twice the night before surgery and within 2-3 hours before surgery. The entire drink is meant to be consumed within 15 minutes.
  Interventions: Drug: Maltodextrin solution
- Placebo Group (Placebo Comparator): Patients in the intervention group will receive a placebo in 400 millilitres (mL) of water twice the night before surgery and within 2-3 hours before surgery. The entire drink is meant to be consumed within 15 minutes.
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: Maltodextrin solution — The oral preparation of 50 grams of Maltodextrin solution mixed in 400 mL of water
  Other Names: Intervention group
  Arms: Intervention Group
Drug: Placebo solution — Specifically formulated placebo to provide a similar taste and texture to Maltodextrin, without the same carbohydrate characteristics
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
A randomized, controlled, double-blinded clinical trial evaluating the effect of the administration of a Maltodextrin solution on cardiac function in patients presenting for coronary artery bypass grafting surgery with a reduced left ventricular ejection fraction.

DETAILED DESCRIPTION:
This randomized, double-blinded clinical trial will test the primary hypothesis that patients receiving preoperative maltodextrin will have an improved intraoperative left ventricular ejection fraction (LVEF), as measured by three-dimensional echocardiography, compared to patients who receive a placebo drink. Seventy patients will be recruited and randomized to each group in a 1:1 ratio.

The second hypothesis is that administering preoperative Maltodextrin to cardiac surgery patients enhances the quality of recovery, as measured by the Quality of Recovery-15 score. Each patient will undergo this questionnaire 48 hours after surgery.

The third hypothesis is that Maltodextrin improves cardiac function by its effect on myocardial glycogen content. This will be evaluated in two ways. First, a separate group of 20 patients will undergo the hyperinsulinemic-normoglycemic clamp (HNC) to have a high-insulin level during surgery with these patients randomized to Maltodextrin or placebo. In addition, 20 patients from the main study will undergo myocardial biopsies to assess the glycogen content in the Maltodextrin and the placebo groups.

Pre-defined subgroups:

* Need for vasopressors or inotropes during measures of cardiac function vs no need
* Male versus female
* Diabetic versus non-diabetic
* Sarcopenic versus non-sarcopenic
* Malnourished versus non-malnourished

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Presenting for coronary artery bypass grafting surgery
* Preoperative left ventricular ejection fraction < 50%
* First case of the day (7:30am start time)

Exclusion Criteria:

* Dysphagia, gastroparesis
* Cannot tolerate oral intake
* Celiac disease
* Type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative three-dimensional left ventricular ejection fraction (3-D LVEF) | After induction of anesthesia, prior to the start of surgery, and at the conclusion of surgery, just after chest closure
  LVEF as measured from a 3-D dataset

SECONDARY OUTCOMES:
Right Ventricular 3-D EF | After induction of anesthesia, prior to the start of surgery, and at the conclusion of surgery, just after chest closure
  Right ventricular ejection fraction as measured from a 3-D dataset
Left Ventricular Strain | After induction of anesthesia, prior to the start of surgery, and at the conclusion of surgery, just after chest closure
  Strain values obtain by left ventricular speckle tracking
E/e' ratio | After induction of anesthesia, prior to the start of surgery, and at the conclusion of surgery, just after chest closure
  early diastolic mitral inflow velocity to early diastolic mitral annulus velocity
Cardiac Index | After induction of anesthesia, prior to the start of surgery, and at the conclusion of surgery, just after chest closure
  Cardiac index, defined as cardiac output / body surface area, as measured by pulmonary artery catheter
Vasopressors and Inotrope Use | First 1-7 days after surgery
  Dose of vasopressors and inotropes used upon arrival to ICU, and the length of time that they were used
Time to extubation | First 1-48 hours after surgery
  Time from ICU arrival to extubation
Hyperglycemia | First 1-48 hours after surgery
  Incidence of glucose levels greater than 10mmol/L
Insulin Requirements | First 1-48 hours after surgery
  Dose of insulin required after surgery
Length of ICU stay | First 1-7 days after surgery
  Time from surgery to ICU discharge
Hospital Length of Stay | 1-4 weeks after surgery
  Time from surgery to discharge from the hospital
Postoperative complications | 1-4 weeks after surgery
  as death, need for intra aortic balloon pump, dialysis, stroke, positive bacterial culture from the wound or blood
Quality of Recovery | At 48 hours after surgery
  Quality of Recovery after surgery as measured by the QoR-15 questionnaire
Hyperinsulinemic-normoglycemic clamp (HNC) details | During the surgery
  Total dose of insulin and glucose needed, and the peak insulin dose required
Myocardial glycogen content | From biopsies optained intraoperatively, during cardiopulmonary bypass
  Measurements of myocardial mitochondrial function

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cameron, MDCM, MPH, Principal Investigator — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada